CLINICAL TRIAL: NCT04203134
Title: Protective Mouth Guards in Burning Mouth Syndrome (Prospective Study)
Brief Title: Burning Mouth Syndrome Mouth Guard Prospective Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB201902692; OCR29702 (Other: University of Florida)
Record Dates: First submitted 2019-12-16; First posted 2019-12-18 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Burning Mouth Syndrome; Burning Mouth
MeSH Terms: conditions — Burning Mouth Syndrome | interventions — Mouth Protectors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Patients in the randomly assigned treatment group will receive a mouthguard at first visit along with standard treatment of BMS.
  Interventions: Device: Mouthguard
- Control Group (No Intervention): Control group will proceed through treatment for BMS in an otherwise standard treatment protocol and will not receive a mouthguard.

INTERVENTIONS:
Device: Mouthguard — The mouthguard is a thin clear acrylic protector fabricated from an impression of a patient's upper teeth and palate. The acrylic protector will be trimmed and will fit onto the patient's upper teeth and palate for use during the day, except when eating to minimize trauma to the tongue that exacerbates burning tongue pain.
  Arms: Treatment Group

SUMMARY:
This study will seek to test the effectiveness of a nonpharmacologic therapy for burning mouth syndrome (BMS). This nonpharmacologic therapy approach will be the fabrication a protective acrylic mouthguard for the maxillary arch and palate.

DETAILED DESCRIPTION:
The study involves a nonpharmacologic and non-invasive treatment method for BMS which will be administered randomly (flipping a coin) to half of the study subjects, (case group) in addition to normal condition treatment protocol for BMS.

ELIGIBILITY:
Inclusion Criteria:

• New patients diagnosed with BMS seen in the oral medicine clinic for the study period.

Exclusion criteria includes:

• Patients with inconclusive diagnosis or evidence of underlying condition that may be causing oral burning therefore excluding BMS as a diagnosis

Inclusion Criteria:

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2021-06-18 (Actual); Study Completion 2021-06-18 (Actual)

PRIMARY OUTCOMES:
Effectiveness in pain control | Baseline through 6 month
  patient reported pain level using self reported word descriptor scale. Range from 0 - 5, with 0 as "no pain" and 5 as "excruciating pain"

CONTACTS AND LOCATIONS:
Overall Officials: Austin Belknap, Principal Investigator — University of Florida
Locations (1):
- University of Florida College of Dentistry, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No